CLINICAL TRIAL: NCT06585488
Title: A Phase 1a/1b Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BGB-53038, a Pan-KRAS Inhibitor, as Monotherapy or in Combinations in Patients With Advanced or Metastatic Solid Tumors With KRAS Mutations or Amplifications
Brief Title: A First-in-human Study of BGB-53038, a Pan-KRAS Inhibitor, Alone or in Combinations in Participants With Advanced or Metastatic Solid Tumors With KRAS Mutations or Amplification
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-53038-101; 2024-514704-13-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Solid Tumors; Advanced Non-squamous Non-small-cell Lung Cancer; Advanced Colorectal Cancer; Advanced Pancreatic Ductal Adenocarcinoma; Advanced Gastric Cancer; Advanced Gastroesophageal Junction Cancer; Advanced Esophageal Adenocarcinoma
Keywords: KRAS wild type amplification; Metastatic Solid Tumors; Advanced Non-squamous Non-small-cell Lung Cancer; Advanced Colorectal Cancer; Advanced Pancreatic Ductal Adenocarcinoma; Advanced Gastric Cancer; Advanced Gastroesophageal Junction Cancer; Advanced Esophageal Adenocarcinoma
MeSH Terms: interventions — tislelizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1a: Part A (Monotherapy Dose Escalation) (Experimental): Sequential cohorts will be evaluated to determine the Recommended Dose for Expansion (RDFE) of BGB-53038 as a monotherapy.
  Interventions: Drug: BGB-53038
- Phase 1a: Part B (Monotherapy Safety Expansion) (Experimental): Participants will be enrolled at dose levels determined in Part A with the Safety Monitoring Committee to confirm the final RDFE(s) for BGB-53038 monotherapy.
  Interventions: Drug: BGB-53038
- Phase 1a: Part C (Combination Therapy Dose Escalation) (Experimental): Sequential cohorts with increasing doses will be evaluated to determine the RDFE(s) for BGB-53038 in combination with tislelizumab or cetuximab.
  Interventions: Drug: BGB-53038; Drug: Tislelizumab; Drug: Cetuximab
- Phase 1b: Part D (Monotherapy Dose Expansion) (Experimental): Participants will be enrolled to receive the RDFE(s) of BGB-53038 monotherapy
  Interventions: Drug: BGB-53038
- Phase 1b: Part E (Combination Therapy Dose Expansion) (Experimental): Participants will be enrolled to receive BGB-53038 at the RDFE(s) as determined in Part C of Phase 1a in combination with tislelizumab and in combination with cetuximab, respectively.
  Interventions: Drug: BGB-53038; Drug: Tislelizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: BGB-53038 — Administered orally
Drug: Tislelizumab — administered by intravenous infusion
  Other Names: Tevimbra
  Arms: Phase 1a: Part C (Combination Therapy Dose Escalation); Phase 1b: Part E (Combination Therapy Dose Expansion)
Drug: Cetuximab — administered by intravenous infusion
  Arms: Phase 1a: Part C (Combination Therapy Dose Escalation); Phase 1b: Part E (Combination Therapy Dose Expansion)

SUMMARY:
This is a first-in-human (FIH), open-label, multicenter, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BGB-53038 as monotherapy in participants with advanced or metastatic solid tumors harboring KRAS mutations or amplification, as well as when used in combination with tislelizumab (also known as BGB-A317) in participants with nonsquamous non-small cell lung cancer (NSCLC) and used in combination with cetuximab in participants with colorectal cancer (CRC). The study consists of 2 phases: Phase 1a Dose Escalation and Safety Expansion and Phase 1b Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Must sign a written ICF; and understand and agree to comply with the requirements of the study and the schedule of activities.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
3. Participants must have evidence of a KRAS mutation or wild-type amplification (copy number ≥ 8) based on testing of either tumor tissue or liquid biopsy (blood or plasma) as determined by local laboratory
4. Able to provide an archived tumor tissue sample or fresh biopsy sample.
5. ≥ 1 measurable lesion per RECIST v1.1.
6. Adequate organ function.
7. Females of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, for > 7 days after the last dose of BGB-53038, > 120 days after the last dose of tislelizumab, or > 2 months after the last dose of cetuximab, whichever is later
8. Nonsterile males must be willing to use a highly effective method of birth control for the duration of the study treatment period and for ≥ 4 months after the last dose of study drug(s).

Exclusion Criteria:

1. Participants with tumors harboring KRAS G12R mutation.
2. Participants who have prior therapy with other anti-RAS treatment, including, but not limited to, therapy targeting specific KRAS allele mutation inhibitors, pan-KRAS inhibitors, and other pan-RAS inhibitors
3. Participants with active leptomeningeal disease or uncontrolled, untreated brain metastasis. Participants with a history of treated and, at the time of screening, stable CNS metastases are eligible, provided they meet select criteria.
4. Any malignancy ≤ 2 years before the first dose of study treatment(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast).
5. Participants with untreated chronic hepatitis B or chronic HBV carriers with HBV DNA ≥ 500 IU/mL (or ≥ 2500 copies/mL) at screening. Participants with active hepatitis C.
6. Participants with clinically significant infections (including tuberculosis infection) requiring systemic (oral or intravenous) antibacterial, antifungal, or antiviral therapy ≤ 14 days before the first dose of study treatment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 2 years
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) characterized by type, frequency, severity (as graded by the National Cancer Institute-Common Terminology Criteria for Adverse Events [NCICTCAE] Version [v] 5.0), timing, seriousness, and relationship to study drug(s); and adverse events meeting protocol-defined dose-limiting toxicity (DLT) criteria
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-53038 | Up to approximately 2 years
  defined as the highest dose at which 30% of the participants experienced a DLT or the highest dose administered, respectively.
Phase 1a: Recommended Dose for Expansion (RDFE) of BGB-53038 | Up to approximately 2 years
  The potential RDFE(s) of BGB-53038 as monotherapy or in combination with other antitumor therapies (tislelizumab or cetuximab) will be determined based on the totality of safety, tolerability, pharmacokinetics (PK), pharmacodynamics, preliminary antitumor activity, and any other relevant data, as available.
Phase 1b: Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator using RECIST v1.1
Phase 1b: Recommended Phase 2 Dose (RP2D) of BGB-53038 | Up to approximately 2 years
  The RP2D of BGB-53038 as monotherapy or in combination with other antitumor therapies (tislelizumab or cetuximab) will be determined based on safety, long-term tolerability, PK, preliminary antitumor activity, and any other relevant data, as available

SECONDARY OUTCOMES:
Phase 1a: Single-dose and steady-state area under the concentration-time curve (AUC) of BGB-53038 | Up to approximately 2 years
Phase 1a: Single-dose and steady-state Half-life (t1/2) of BGB-53038 | Up to approximately 2 years
Phase 1a: Single-dose and steady-state maximum observed plasma concentration (Cmax) of BGB-53038 | Up to approximately 2 years
Phase 1a: Single-dose and steady-state trough concentration (Ctrough) of BGB-53038 | Up to approximately 2 years
Phase 1b: ORR | Up to approximately 2 years
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) assessed by the investigator using RECIST v1.1.
Duration of Response (DOR) | Up to approximately 2 years
  DOR is defined as the time from the first determination of an objective response per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first as assessed by the investigator.
Time to Response (TRR) | Up to approximately 2 years
  defined as the time from the date of first dose of study drug to first documentation of response as assessed by the investigator per RECIST v1.1
Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the percentage of participants who achieve CR, PR, or stable disease (SD) lasting ≥ 24 weeks as assessed by the investigator per RECIST v1.1
Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of the first dose of study drug(s) to the date of the first documentation of progressive disease assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1b: Overall Survival (OS) | Up to approximately 2 years
  defined as the time from the date of first dose of study drug until the date of death from any cause
Phase 1b: Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 2 years
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) characterized by type, frequency, severity (as graded by the NCI-CTCAE v5.0), timing, seriousness, and relationship to study drug(s)
Plasma concentrations of BGB-53038 | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (18):
- United States (4):
  - Usc Norris Comprehensive Cancer Center (Nccc), Los Angeles, California
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Sidney Kimmel Comprehensive Cancer At Johns Hopkins, Baltimore, Maryland
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Monash Health, Clayton, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (3):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
- Auckland City Hospital, Auckland, New Zealand
- South Korea (5):
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
- Start Madrid Fundacion Jimenez Diaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/